CLINICAL TRIAL: NCT03242005
Title: The PSIQS Study - User Experience With the Pro-Set Over Intended Wear of 3 Days With New Instructions and Requirement to be Inserted With the Quick-Serter
Brief Title: The PSIQS Study - User Experience With Pro-Set
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision to not proceed with study - no subjects enrolled
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DBC-17SCARL23
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Pro-set® vs. Quick-set® (Experimental): Subjects will be randomized to start with one of the study subcutaneous insulin administration sets (MiniMed® Pro-set® or MiniMed® Quick-set®). After completing the first study period,subjects will be placed in the alternative group according to the cross-over study design.
  Interventions: Device: MiniMed® Pro-set®; Device: MiniMed® Quick-set®

INTERVENTIONS:
Device: MiniMed® Pro-set® — Utilization of the MiniMed® Pro-set® to administer the subject's current insulin therapy.
Device: MiniMed® Quick-set® — Utilization of the MiniMed® Quick-set® to administer the subject's current insulin therapy.

SUMMARY:
Open label, randomized 2-period cross-over study comparing two continuous subcutaneous insulin infusion sets ; MiniMed® Pro-set® with BD FlowSmart™ technology and MiniMed® Quick-set®

ELIGIBILITY:
Inclusion Criteria:

* Must be between 13 and 70 years of age (inclusive)
* Must have been previously diagnosed with type 1 diabetes mellitus
* Must be using one of the following Medtronic insulin pumps with the Paradigm connector (note 670G excluded) for at least 6 months prior to enrollment. These pumps must have the ability to upload data to Medtronic CareLink Therapy Management software.

  1. MiniMed Paradigm Revel™ Insulin Pump - models 523 (1.8 mL reservoir) and 723 (3 mL reservoir)
  2. MiniMed 530G Pump - models 551 (1.8 mL reservoir) and 751 (3 mL reservoir)
  3. MiniMed 630G System
* Must have been using the Medtronic Enlite CGM for at least 3 months prior to enrollment, and are currently doing so
* Must routinely insert their own infusion set (may be inserted manually or with an inserter or with an integrated set/inserter, i.e. Mio)
* If instructed, must be willing to insert all assigned infusion sets with a mechanical inserter
* Must have another form of insulin delivery available (i.e. vial and syringe or pen and pen needle)
* Must agree to continue using current Medtronic Enlite CGM throughout the study
* Willing to have insulin pump, BGM and CGM data downloaded into Medtronic CareLink Therapy Management Software (requires subject CareLink logon ID and password)
* In stable health status with no acute or significant illness, in the opinion of the investigator or designee
* Able to read, write and follow instructions in English
* Able and willing to provide informed consent
* Able and willing to comply with study procedures

Exclusion Criteria:

* Pregnant (self-attestation) or nursing
* Currently using a body-worn patch insulin infusion pump, e.g. Omnipod or V-Go
* Currently using the Medtronic Model 670G pump and associated CGM
* Current or past participation in previous BD Study DBC-16SCARL21
* History of bleeding disorder or easy bruising.
* Currently taking anti-platelet therapy or anticoagulants (use of up to 81 mg per day of aspirin is permitted).
* Known blood borne infections.
* History of recurrent dermatological condition or skin disorder (e.g. psoriasis, eczema, pre-existing dermatitis).
* Skin abnormalities, anomalies or conditions (e.g. sunburn, tattoos, extensive scarring, lipohypertrophy) located at or very close to the intended insertion site.
* Physical condition that restricts dexterity and may limit ability to perform study procedures (i.e. severe neuropathy or arthritis of the hands; self-reported)
* Currently participating in any other clinical investigation that conflicts with this study
* Employed by, or currently serving as a contractor or consultant to BD, Medtronic or study site
* Any other condition the investigator or designee deems to pose an unacceptable risk to the subject in the study

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Compare Pro-set® vs. Quick-set® for non-inferiority for set insertion failures (set removal) due to either occlusion alerts or hyperglycemia | 6 hours from time of insertion

SECONDARY OUTCOMES:
Compare Pro-set® vs. Quick-set® for set removals due to hyperglycemia; > 400mg/dl. | 6 hours from time of insertion
Compare Pro-set® vs. Quick- set® for set removals due to set failure; hyperglycemia >250mg/dl. | 72 hours of set wear that occurs at 6 hours or later after insertion
Compare Pro-set® vs. Quick- set® for set removals at less than 60 hours post insertion. | 60 hours post insertion
Compare Pro-set® vs. Quick- set® for duration of wear | % reaching 12 hours, % reaching 24 hours, % reaching 36 hours, % reaching 48 hours, % reaching 60 hours, and % reaching 72 hours)

IPD SHARING:
Plan to Share IPD: No